CLINICAL TRIAL: NCT00279643
Title: The Effect of Laser Hair Removal on Markers of Follicular Stem Cells
Brief Title: The Effect of Laser Hair Removal on Permanent Hair Reduction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey S. Orringer, Professor of Dermatology, Medical School, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Derm 543
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Laser Hair Removal in Healthy Subjects
Keywords: Laser; immunohistochemical staining; Laser Hair Removal; follicular stem cells; keratin 15

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Laser Hair Removal

SUMMARY:
The purpose of this study is to learn more about how hair removal with lasers achieves, what appears to be, permanent hair reduction. Laser hair removal has become one of the most popular and commonly performed procedures in cosmetic dermatology. However, relatively little is known about how the permanent reduction in the treated areas occurs. Recently, it has been discovered that certain cells in the hair follicle must be destroyed in order to achieve permanent hair reduction. A marker of these types of cells known as keratin 15 has been identified. By measuring the amount of keratin 15 before and after laser therapy, we hope to gain a better understanding of how lasers cause hair reduction on a biochemical level.

DETAILED DESCRIPTION:
Laser hair removal has become one of the most popular and commonly performed procedures in cosmetic dermatology. However, relatively little is known about the mechanisms involved in achieving what clinically appears to be permanent reduction in hair density in treated areas. We postulate that in order to achieve permanent hair reduction, stem cells located in the bulge region of the follicle must be destroyed. Recently, a marker of follicular stem cells (keratin 15) has been identified and noted to be detectable using immunohistochemical techniques. In addition, several other immunohistochemical markers for various components of the hair follicle are available.

We propose to quantitatively measure the effects of laser hair removal on the immunohistochemical staining properties of treated follicles with respect to keratin 15 and other follicular markers. We hypothesize that the degree of such staining will be greatly reduced following laser therapy, thus providing, to our knowledge, the first biochemical evidence to support permanence of the treatment's effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older of either gender.
2. At least moderately dense axillary (armpit) hair that is dark (not blonde or white) in color.
3. Subjects must understand and sign the informed consent documents prior to participation.
4. Subjects must be in generally good health.
5. Subjects must be willing and able to comply with the requirements of the protocol
6. You must live within a reasonable driving distance of Ann Arbor, Michigan, and/or be able to attend all of the scheduled appointments during the study.

Exclusion Criteria:

1. Oral retinoid use within one year of study entry.
2. History of prior laser therapy or electrolysis of the axillae.
3. Subjects who do not desire permanent reduction in axillary hair.
4. Non-compliant subjects.
5. Pregnant or nursing subjects.
6. Subjects with a significant medical history or concurrent illness/condition that the investigator(s) feel is not safe for study participation.
7. Active infection of the site to be treated or a history of herpes simplex or zoster infection at the site to be treated.
8. History of keloid scar formation.
9. Known history of allergy or sensitivity to lidocaine.
10. History of waxing, plucking, or bleaching of the hair for 6 weeks prior to the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-01; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
measurement of the effects of laser hair removal on the immunohistochemical staining properties of human hair follicles, including the putative stem cells of the bulge region.

SECONDARY OUTCOMES:
Hair Removal

CONTACTS AND LOCATIONS:
Overall Officials: John J Voorhees, MD, Study Chair — University of Michigan
Locations (1):
- University of Michigan Department of Dermatology, Ann Arbor, Michigan, United States